CLINICAL TRIAL: NCT01641939
Title: A Randomized, Multicenter, Adaptive Phase II/III Study To Evaluate The Efficacy And Safety Of Trastuzumab Emtansine (T-DM1) Versus Taxane (Docetaxel Or Paclitaxel) In Patients With Previously Treated Locally Advanced Or Metastatic HER2-Positive Gastric Cancer, Including Adenocarcinoma Of The Gastroesophageal Junction
Brief Title: A Study of Trastuzumab Emtansine Versus Taxane in Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Advanced Gastric Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO27952; 2012-000660-22 (EudraCT Number)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — taxane; Ado-Trastuzumab Emtansine

ARMS (3):
- Standard taxane therapy (Active Comparator): Docetaxel will be administered at 75 milligram per meter square (mg/m^2) intravenous (IV) on Day 1 of a 21-day cycle, or paclitaxel will administered at 80 mg/m^2 IV weekly (Days 1, 8, and 15 of a 21 day cycle) according to investigator choice until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
  Interventions: Drug: Taxane
- trastuzumab emtansine 2.4 mg (Experimental): Trastuzumab emtansine will be administered on Day 1, 8, and 15 of a 21-day cycle at 2.4 mg/kg IV infusion until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
  Interventions: Drug: trastuzumab emtansine
- trastuzumab emtansine 3.6 mg (Experimental): Trastuzumab emtansine will be administered on Day 1 of a 21-day cycle at 3.6 mg/kg IV infusion until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
  Interventions: Drug: trastuzumab emtansine

INTERVENTIONS:
Drug: Taxane — Standard taxane (docetaxel 75 mg/m^2 IV every 3 weeks or paclitaxel 80 mg/m^2) IV once a week according to investigator choice.
  Arms: Standard taxane therapy
Drug: trastuzumab emtansine — trastuzumab emtansine 3.6 mg/kg IV every 3 weeks
  Arms: trastuzumab emtansine 3.6 mg
Drug: trastuzumab emtansine — trastuzumab emtansine 2.4 mg/kg IV once a week
  Arms: trastuzumab emtansine 2.4 mg

SUMMARY:
This multicenter, randomized, adaptive Phase II/III study will evaluate the efficacy and safety of trastuzumab emtansine (T-DM1) compared to standard taxane (docetaxel or paclitaxel) treatment in participants with human epidermal growth factor receptor 2 (HER2)-positive advanced gastric cancer. At the start of the trial (stage 1), participants will be randomized with a ratio 2:2:1 to one of three treatment arms: Arm A: trastuzumab emtansine 3.6 milligram per kilogram (mg/kg) per intravenous injection (IV) every 3 weeks; Arm B: trastuzumab emtansine 2.4 mg/kg IV every week; Arm C: standard taxane therapy (docetaxel 75 milligram per meter square [mg/m^2] IV every 3 weeks or paclitaxel 80 mg/m^2 kg IV every week per investigator choice). At the end of the first stage of the study, the dose and schedule of trastuzumab emtansine that will be used in the second stage of the study will be selected by an Independent Data Monitoring Committee (IDMC). The regimen selection analysis will be made after approximately 100 participants across all three study arms have been treated for at least 12 weeks.

Once a trastuzumab emtansine regimen has been selected, Stage I participants who were assigned to the treatment arm which was selected for Stage II of the study and participants who were in the standard taxane group will continue to receive their assigned treatment regimen. Stage I participants who were assigned to the regimen that was not selected for further evaluation will continue to receive their assigned regimen and will continue to be followed for efficacy and safety. In Stage II of the study, additional participants will be recruited and randomized with a ratio 2:1 to either the selected regimen of trastuzumab emtansine or to the standard taxane therapy. Participants will receive study treatment until disease progression, unacceptable toxicity, initiation of another cancer therapy or withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 12 weeks from the first dose of study treatment
* Measurable and/or evaluable disease based on Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* Adequate organ function as determined by the following laboratory results, within 28 days prior to randomization
* Participants must have a history of advanced gastric cancer (AGC), defined as unresectable and locally advanced or metastatic gastric cancer, including adenocarcinoma of the gastroesophageal junction (GEJ), and must have experienced disease progression during or after first-line therapy for their disease
* HER2-positive tumor (primary tumor or metastatic lesion) as confirmed by central laboratory HER2 testing (immunohistochemistry and/or in-situ hybridization)
* Participants must have received at least one prior chemotherapy regimen for AGC; prior therapy does not need to have included HER2-directed therapy.
* First-line therapy for AGC, including adenocarcinoma of the GEJ, must have included a combination of at least a platinum- and a fluoropyrimidine-based treatment given concurrently; prior therapy does not need to have included a HER2-directed therapy.
* Adjuvant or neoadjuvant therapy for AGC is allowed.

Exclusion Criteria:

* An interval shorter than 21 days from the last dose of chemotherapy or HER2-directed therapy until the time of randomization
* Prior treatment with trastuzumab emtansine, docetaxel, or paclitaxel either as single agents or as part of a treatment regimen.
* Treatment with any investigational anticancer drug within 21 days of the first study treatment administration
* More than one prior line of therapy for advanced gastric cancer
* History of other malignancy within the previous 5 years except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other malignancies with an expected curative outcome
* Brain metastases that are untreated or symptomatic or require any radiation, surgery, or steroid therapy to control symptoms from brain metastases within 1 month of randomization
* Peripheral neuropathy Grade >/=2
* Uncontrolled cardiopulmonary dysfunction (e.g., high blood pressure, serious cardiac arrhythmia)
* Other current, severe, uncontrolled systemic disease (e.g., clinically significant metabolic disease, wound healing disorders, ulcers)
* Clinically significant bleeding within 30 days before enrollment
* For female participants, current pregnancy or lactation
* Major surgical procedure or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* Infection with Human immunodeficiency virus (HIV) or hepatitis B virus, hepatitis C virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2012-09-03 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (148):
- United States (10):
  - Comprehensive Blood/Cancer Ctr, Bakersfield, California
  - Stanford University School of Medicine, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Kansas; Medical Center & Medical pavilion, Westwood, Kansas
  - Norton Healthcare Inc., Louisville, Kentucky
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Vanderbilt, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Argentina (3):
  - Fundación Investigar, Buenos Aires
  - Hospital de Gastroenterologia Dr. Bonorino Udaondo ; Servicio de Oncología, Buenos Aires
  - Instituto de Oncología de Rosario, Rosario
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (7):
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
- Canada (4):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Brampton Memorial Hospital, William Osler Health Center, Brampton, Ontario
  - Toronto East General Hospital; Haematology/Oncology, Toronto, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
- China (20):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - the First Hospital of Jilin University, Changchun
  - Changzhou First People's Hospital, Changzhou
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - The 81st Hospital of P.L.A., Nanjing
  - Affiliated Hospital of Nantong University, Nantong
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - General Hospital of Shenyang Military Command of PLA, Shenyang
  - Union Hospital of Tongji Medical College, Dept. of Cancer Center; Cancer Center, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Fakultní Nemocnice V Motole; Radioterapeuticko-Onkologicke Oddeleni, Prague
- Tampere University Hospital; Dept of Oncology, Tampere, Finland
- France (7):
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Hopital Beaujon; Gastro Enterologie 1, Clichy
  - Centre Val Aurelle Paul Lamarque; Medecine A1 A2, Montpellier
  - Hopital Saint Antoine; Hepatologie-Gastr-Enterologie, Paris
  - Hop Europeen Georges Pompidou; Gastro Enterologie, Paris
  - Hopital Robert Debre; Gastro Enterologie, Reims
  - Hopital Purpan; Unite Onco Digestive, Toulouse
- Germany (6):
  - Charité-Universitätsm. Berlin; Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunolo., Berlin
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum "Carl Gustav Carus"; Med. Klinik & Poliklinik I, Arbeitsgr. intern. Onkologie, Dresden
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - Tagesklinik Landshut; Hämatologie/Onkologie, Landshut
  - Onkologische Gemeinschaftspraxis, Magdeburg
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hungary (4):
  - Fovarosi Szent Laszlo Korhaz-Rendelointezet; Onkologiai Osztaly X, Budapest
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Hetenyi Geza County Hospital; Onkologiai Kozpont, Szolnok
  - Zala Megyei Kórház, Külsö Kórház, Pózva; Onkológiai Osztály, Zalaegerszeg
- Italy (5):
  - Campus Universitario S.Venuta; Centro Oncologico T.Campanella, Catanzaro, Calabria
  - AZ.Osp S. Orsola - Malpighi-Reparto di Oncologia Medica, Bologna, Emilia-Romagna
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - A.O. Universitaria Pisana; Oncologia, Pisa, Tuscany
- Japan (19):
  - Aichi Cancer Center Hospital; Clinical Oncology, Aichi
  - Chiba Cancer Center; Gastroenterology, Chiba
  - National Cancer Center Hospital East; Gastroenterology, Chiba
  - National Hospital Organization Shikoku Cancer Center; Gastroenterology, Ehime
  - Hokkaido University Hospital：Gastroenterology, Hokkaido
  - Hyogo College Of Medicine; Upper Gastroenterology, Hyōgo
  - Hyogo Cancer Center; Gastroenterology, Hyōgo
  - Ibaraki Prefectural Central Hospital; Gastroenterology, Ibaraki
  - Tohoku Uni Hospital; Clinical Oncology, Miyagi
  - Osaka University Hospital; Surgery, Osaka
  - Kindai University Hospital; Medical Oncology, Osaka
  - Saitama Cancer Center; Gastroenterology, Saitama
  - Shizuoka Cancer Center; Gastroenterology, Shizuoka
  - Shizuoka General Hospital; Clinical Oncology, Shizuoka
  - Tochigi Cancer Center; Medical Oncology, Tochigi
  - National Cancer Center Hospital; Gastrointestinal Oncology, Tokyo
  - Toranomon Hospital; Medical Oncology, Tokyo
  - Tokyo Metropolitan Komagome Hospital; Chemotherapy, Tokyo
  - The Cancer Institute Hospital, JFCR; Gastroenterology, Tokyo
- Malaysia (2):
  - Hospital Wanita dan Kanak-Kanak Sabah, Sabah, Sabah
  - University Malaya Medical Centre; Clinical Oncology Unit,, Kuala Lumpur
- Mexico (3):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Centro Estatal De Cancerologia De Chihuahua; Servicio De Hematologia Banco De Sangre, Chihuahua City
  - Hospital General de México; Unidad de Oncologia, Mexico City
- Centro Hemato Oncologico Paitilla, Panama City, Panama
- Peru (4):
  - Hospital Nacional Almanzor Aguinaga Asenjo; Unidad De Investigacion Del Servicio De Oncologia Medica, Chiclayo
  - Hospital Nacional Adolfo Guevara Velasco, Cusco
  - Hospital Nacional Edgardo Rebagliati Martins, Jesus Maria
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
- Philippines (2):
  - Perpetual Succour Hospital, Cebu
  - Veterans Memorial Medical Ctr; Cancer Research Centre, Quezon City, Luzon
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wielkopolskie Centrum Onkologii; im. Marii Skłodowskiej-Curie, Poznan
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
  - Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie; Klinika Gastroenterologii Onkologicznej, Warsaw
- Romania (4):
  - Institutul Clinic Fundeni Bucuresti, Bucharest
  - Spitalul Universitar CF Cluj-Napoca; Sectia Oncologie, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Spitalul Clinic Judetean Mures; Oncologie Medicala, Târgu Mureş
- Russia (5):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Omsk Region Clinical Oncology Dispensary; 1St Sergical Department, Omsk
  - State Budget Institution of Healthcare of Stavropol region Pyatigorsk Oncology Dispensary, Pyatigorsk
  - Tula Regional Oncology Dispensary, Tula
- National Cancer Centre, Singapore, Singapore
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center; Medical Oncology, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Korea University Anam Hospital; Oncology Haemotology, Seoul
  - Seoul St.Mary's Hospital; Medical Oncology, Seoul
- Spain (8):
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, La Coruña
  - Hospital Univ. Central de Asturias; Servicio de Oncologia, Oviedo, Principality of Asturias
  - Hospital Clinic i Provincial; Servicio de Farmacia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital; Dept of Hem and Onc, Kaohsung
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Chang Gung Medical Foundation - Linkou; Division of Hematology- Oncology, Taoyuan District
- Turkey (Türkiye) (5):
  - Ataturk University Medical Faculty Yakutiye Research Hospital Medical Oncology Department, Erzurum
  - Istanbul Bilim University School Of Medicine; Department Of Medical Oncology, Istanbul
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Ege Uni Medical Faculty; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara
- United Kingdom (6):
  - Velindre Cancer Centre; Oncology Dept, Cardiff
  - The Beatson West of Scotland Cancer Centre; Cancer Clinical Trials Unit, Glasgow
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - BRISTOL ONCOLOGY CENTRE; CLINICAL TRIALS UNIT; R & D department, Weston-super-Mare

REFERENCES:
- [Derived] Shah MA, Kang YK, Thuss-Patience PC, Ohtsu A, Ajani JA, Van Cutsem E, Hoersch S, Harle-Yge ML, de Haas SL. Biomarker analysis of the GATSBY study of trastuzumab emtansine versus a taxane in previously treated HER2-positive advanced gastric/gastroesophageal junction cancer. Gastric Cancer. 2019 Jul;22(4):803-816. doi: 10.1007/s10120-018-00923-7. Epub 2019 Jan 31. PMID 30706247
- [Derived] Thuss-Patience PC, Shah MA, Ohtsu A, Van Cutsem E, Ajani JA, Castro H, Mansoor W, Chung HC, Bodoky G, Shitara K, Phillips GDL, van der Horst T, Harle-Yge ML, Althaus BL, Kang YK. Trastuzumab emtansine versus taxane use for previously treated HER2-positive locally advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma (GATSBY): an international randomised, open-label, adaptive, phase 2/3 study. Lancet Oncol. 2017 May;18(5):640-653. doi: 10.1016/S1470-2045(17)30111-0. Epub 2017 Mar 23. PMID 28343975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 415 participants were randomized, of these 117 participants in taxane arm, 228 participants in 2.4 milligram per kilogram (mg/kg) trastuzumab emtansine arm, and 70 participants in 3.6 mg/kg trastuzumab emtansine arm received at least one dose of the treatment.
Groups:
- Standard Taxane Therapy: Docetaxel was administered at 75 milligram per meter square (mg/m^2) intravenously (IV) on Day 1 of a 21-day cycle, or paclitaxel was administered at 80 mg/m^2 IV weekly (Days 1, 8, and 15 of a 21 day cycle) as per investigator's choice, until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
- Trastuzumab Emtansine 2.4 mg: Trastuzumab emtansine was administered on Days 1, 8, and 15 of a 21-day cycle at 2.4 milligram per kilogram (mg/kg) IV infusion until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
- Trastuzumab Emtansine 3.6 mg: Trastuzumab emtansine was administered on Days 1 of a 21-day cycle at 3.6 mg/kg IV infusion until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
Period: Overall Study
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Started | 117 | 228 | 70
Stage 1 | 37 | 75 | 70
Stage 2 | 80 | 153 | 0
Completed | 0 | 0 | 0
Not Completed | 117 | 228 | 70
Not completed — Death | 90 | 187 | 61
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 11 | 5
Not completed — Study Terminated by Sponsor | 10 | 28 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis population included all randomized participants; participants grouped according to the therapy they were randomized to receive.
Groups:
- Standard Taxane Therapy: Docetaxel was administered at 75 mg/m^2 IV on Day 1 of a 21-day cycle, or paclitaxel was administered at 80 mg/m^2 IV weekly (Days 1, 8, and 15 of a 21 day cycle) as per investigator's choice, until progression of disease, intolerable toxicity, initiation of another anticancer therapy, or participants and/or physician decision to discontinue.
- Total: Total of all reporting groups
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg | Total
Number analyzed (Participants) | 117 | 228 | 70 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.3) | 60.5 (10.9) | 61.2 (11.4) | 61.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 51 | 17 | 90
  Male | 95 | 177 | 53 | 325

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)- Phase 3
Description: Overall survival was defined as the time between the date of randomization and date of death due to any cause. Kaplan-Meier estimates were used for analysis. Participants for whom no death was reported prior to an analysis cutoff (30 June 2015) was censored at the latest date before the cutoff in which they were known to be alive. All data from the standard taxane therapy and trastuzumab emtansine 2.4 mg (selected treatment arm) from phase 2 and phase 3 (Stage 2) are combined into phase 3 data, and thus cumulative data are provided within the results presented for phase 3. The confirmatory analyses are restricted to comparisons between the taxane arm and the selected trastuzumab emtansine arm (2.4 mg).
Time Frame: Date of randomization until death (up to 2 years 3 months)
Population: ITT population included all randomized participants; participants grouped according to the therapy they were randomized to receive.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 117 | 228
months | 8.6 [7.1 to 11.2] | 7.9 [6.7 to 9.5]
Statistical Analysis 1: Comparison: Standard Taxane Therapy vs Trastuzumab Emtansine 2.4 mg; The unstratified Cox proportional hazards model was used to estimate the hazard ratio. The 95% Confidence Interval (CI) for median was computed using the method of Brookmeyer and Crowley. Reference group: Standard Taxane Therapy; Test type: Superiority or Other; p = 0.8589, Log Rank — One sided p-value with correction for interim treatment selection due to adaptive seamless phase design; Log-Rank test, inverse normal combination test; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.87 to 1.60]

2. Primary Outcome: Overall Survival (OS) - Phase 2 (Dose Selection Portion of the Study)
Description: Overall survival was defined as the time between the date of randomization and date of death due to any cause. Kaplan-Meier estimates were used for analysis. Participants for whom no death was reported prior to an analysis cutoff (10 August 2013) was censored at the latest date before the cutoff in which they were known to be alive.
Time Frame: Date of randomization until death (up to 1 year)
Population: Analysis population included all participants that had been enrolled in phase 2 (stage 1) up to a clinical cut-off date of 10 August 2013; participants grouped according to the therapy they were randomized to receive. Here, N (number of participants analyzed)=number of evaluable participants during phase 2 up to 10 August 2013.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 3.6 mg | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 30 | 58 | 64
weeks | 28.0 [24.0 to NA] — The upper limit of the 95% CI could not be calculated due to the large number of censored events. | 23.0 [18.0 to NA] — The upper limit of the 95% CI could not be calculated due to the large number of censored events. | 36.3 [23.0 to NA] — The upper limit of the 95% CI could not be calculated due to the large number of censored events.
Statistical Analysis 1: Comparison: Standard Taxane Therapy vs Trastuzumab Emtansine 2.4 mg; The unstratified Cox proportional hazards model was used to estimate the hazard ratio. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Reference group: Standard Taxane Therapy; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.32 to 2.03]
Statistical Analysis 2: Comparison: Standard Taxane Therapy vs Trastuzumab Emtansine 3.6 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [0.82 to 4.92]
Statistical Analysis 3: Comparison: Trastuzumab Emtansine 3.6 mg vs Trastuzumab Emtansine 2.4 mg; The unstratified Cox proportional hazards model was used to estimate the hazard ratio. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Reference group: Trastuzumab Emtansine 3.6 mg; Test type: Superiority or Other; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.23 to 0.96]

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST v1.1) - Phase 3
Description: Progressive disease could base on symptom deterioration or was defined as at least a 20 percent (%) increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Tumor assessment was performed using modified RECIST v1.1. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: Date of randomization until disease progression or death, whichever occurred first (assessed at baseline, every 6 weeks up to 2 years 3 months)
Population: as for outcome 1
Measure: Number; unit: percentage participants
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 117 | 228
percentage participants | 88.9 | 93.0

4. Secondary Outcome: Progression Free Survival (PFS) According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST v1.1) - Phase 3
Description: Progression-free survival was defined as the time between the date of randomization and the first date of documented progression or date of death due to any cause, whichever occurred first. Tumor assessment was performed using modified RECIST v1.1. Progressive disease could base on symptom deterioration or was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started or the appearance of one or more new lesions and/or the unequivocal progression of existing non-target lesions. Kaplan-Meier estimates were used for analysis. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure. The confirmatory analyses are restricted to comparisons between the taxane arm and the selected trastuzumab emtansine arm (2.4 mg).
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 117 | 228
months | 2.89 [2.76 to 4.01] | 2.66 [1.61 to 2.79]
Statistical Analysis 1: Comparison: Standard Taxane Therapy vs Trastuzumab Emtansine 2.4 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.308, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.89 to 1.43]

5. Secondary Outcome: Percentage of Participants With Objective Response According to mRECIST v1.1 - Phase 3
Description: Objective response referred to participants with complete response (CR) or partial response (PR). CR: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: greater than or equal to (>=) 30% decrease in sum of the longest diameter (LD) of all target lesions taking as reference the screening sum LD. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments that should have been performed no less than 4 weeks after the criteria for response were first met. Longer intervals as determined by the study protocol were also appropriate. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: as for outcome 3
Population: ITT population included all randomized participants, participants grouped according to the therapy they were randomized to receive. Here, N=number of participants with measurable disease were included in analysis of this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 102 | 204
percentage of participants | 19.6 [12.56 to 28.07] | 20.6 [15.26 to 26.45]

6. Secondary Outcome: Duration of Objective Response (DOR) - Phase 3
Description: DOR: time from the date when a clinical response [CR or PR] was first documented to the date of first documented progressive disease (PD) or death. CR:disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: >= 30% decrease in sum of the LD of all target lesions taking as reference the screening sum LD. PD: could base on symptom deterioration or at least a 20% increase in the sum of diameters of target or non-target lesions and new lesions, taking as reference the smallest sum on study (nadir), including baseline. To be assigned a status of PR or CR, changes in tumor measurements had to be confirmed by repeat assessments that should have been performed no less than 4 weeks after the criteria for response were first met. Longer intervals as determined by the study protocol were also appropriate. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: as for outcome 3
Population: ITT population included all randomized participants, participants grouped according to the therapy they were randomized to receive. Here, N=number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 102 | 204
months | 3.65 [2.76 to 5.55] | 4.27 [3.02 to 6.83]

7. Secondary Outcome: Percentage of Participants With Clinically Significant Improvement in European Organisation for Research and Treatment of Cancer Quality of Life Core Module 30 (EORTC QLQ-C30) Score - Phase 3
Description: The EORTC QLQ-C30 is a validated, cancer-specific 30-item patient-reported measure, and contains 14 domains to assess the impact of cancer treatment on 5 aspects of participants functioning (physical, role, cognitive, emotional, and social), 9 aspects of disease/treatment-related symptoms (fatigue, nausea and vomiting, pain, dyspnea, insomnia, loss of appetite, constipation, diarrhea) and a global QoL/overall health status scale. Questions used 4 point scale (1 'Not at all' to 4 'Very much'; with the exception of the QoL/health status scale which uses a 7-point scale (1 'very poor' to 7 'Excellent'). Each scale is transformed on a scale of 0-100; a higher score equals (=) a better level of functioning or greater degree of symptoms. Change of greater than or equal to (>=) 10-points has been found to be clinically significant. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: Day 1 of each treatment cycle, at the study drug completion visit, and thereafter at follow-up (up to 2 years 3 months)
Population: ITT population included all randomized participants, participants grouped according to the therapy they were randomized to receive. Here, N=number of participants with baseline and at least one post-baseline valid score.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 91 | 189
percentage of participants
  Global Health Status/QoL | 44.0 [33.56 to 54.75] | 34.4 [27.65 to 41.36]
  Appetite loss | 39.6 [29.57 to 50.00] | 30.2 [23.97 to 37.23]
  Cognitive Functioning | 31.9 [22.49 to 42.00] | 28.0 [21.76 to 34.68]
  Constipation | 40.7 [30.48 to 51.47] | 25.9 [19.84 to 32.66]
  Diarrhoea | 23.1 [14.89 to 32.53] | 21.7 [16.23 to 28.15]
  Dyspnea | 19.8 [12.16 to 29.19] | 21.7 [16.23 to 28.15]
  Emotional Functioning | 24.2 [15.98 to 33.56] | 29.1 [22.74 to 35.78]
  Fatigue | 46.2 [36.17 to 56.92] | 40.7 [33.67 to 47.81]
  Nausea/Vomiting | 33.0 [24.04 to 43.08] | 28.0 [21.76 to 34.68]
  Pain | 49.5 [38.80 to 60.14] | 33.9 [27.36 to 40.84]
  Physical Functioning | 17.6 [10.40 to 26.44] | 25.9 [19.84 to 32.66]
  Role Functioning | 29.7 [20.55 to 39.86] | 30.7 [24.20 to 37.75]
  Social Functioning | 34.1 [24.45 to 44.16] | 37.6 [30.80 to 44.48]
  Insomnia | 33.0 [24.04 to 43.08] | 33.3 [26.83 to 40.32]

8. Secondary Outcome: Percentage of Participants With Clinically Significant Improvement in Quality of Life Questionnaire Stomach Cancer Module 22 (QLQ-STO22) Score - Phase 3
Description: The Quality of Life Questionnaire Stomach Cancer Module 22 (QLQ-STO22) supplements the EORTC QLQ-C30 to assess symptoms and treatment-related side effects commonly reported in participants. There are 22 questions which comprise 5 scales (dysphagia, pain, reflux symptom, dietary restrictions, and anxiety) and 4 single items (dry mouth, hair loss, taste, body image). Most questions use 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms. Change of >=10 points has been found to be clinically significant. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: Day 1 of each treatment cycle, at the study drug completion visit, and thereafter at survival follow-up (up to 2 years 3 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 90 | 185
percentage of participants
  Overall | 88.9 [81.15 to 94.54] | 88.1 [82.64 to 92.40]
  Body image | 20.0 [12.31 to 29.33] | 29.7 [23.25 to 36.52]
  Dry Mouth | 30.0 [20.79 to 40.35] | 21.1 [15.44 to 27.28]
  Dietary Restrictions | 41.1 [30.84 to 51.98] | 32.4 [25.75 to 39.66]
  Dysphagia | 35.6 [25.74 to 45.80] | 23.8 [17.84 to 30.31]
  Hair Loss | 11.1 [5.46 to 18.85] | 22.7 [17.07 to 29.29]
  Pain/discomfort | 52.2 [41.43 to 62.45] | 45.4 [38.28 to 52.87]
  Specific Emotional Problems | 63.3 [53.09 to 73.25] | 57.8 [50.71 to 65.05]
  Upper Gastrointestinal Symptoms | 46.7 [36.52 to 57.49] | 42.7 [35.47 to 50.00]

9. Secondary Outcome: Percentage of Participants With Advanced Gastric Cancer (AGC) Symptom Progression - Phase 3
Description: AGC symptomatic progression: a worsening of >=10-points in any 1 of the abdominal discomfort, loss of appetite, weakness and fatigue, upper abdominal pain, change in bowel movement, and/or weight loss scales of the EORTC QLQ-C30 and QLQ-STO22. QLQ-STO22 supplements EORTC QLQ-C30 to assess symptoms and commonly reported treatment-related side effects. There are 22 questions comprise 5 scales (dysphagia, pain, reflux symptom, diet restrictions, anxiety), 4 single items (dry mouth, hair loss, taste, body image), which are related to the symptoms of the disease. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'). All scores and single-items transformed to a scale of 0-100; higher score=better level of functioning or greater degree of symptoms. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: as for outcome 8
Population: ITT population included all randomized participants, participants grouped according to the therapy they were randomized to receive. Here, N=number of participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 117 | 228
percentage of participants | 90.6 | 93.0

10. Secondary Outcome: Time to Advanced Gastric Cancer (AGC) Symptom Progression - Phase 3
Description: Time to AGC symptom were defined as the time from randomization to the first documentation of an increase in at least one of the pre-specified abdominal discomfort, loss of appetite, weakness and fatigue, upper abdominal pain, change in bowel movement, and weight loss subscales of the QLQ STO22 and EORTC QLQ-C30. Cumulative data (up to primary analysis cut-off date of 30-June-2015) are provided for both phase 2 and phase 3 within the results of this measure.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 117 | 228
months | 1.61 [1.41 to 2.17] | 1.51 [1.41 to 1.64]

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Trastuzumab Emtansine (T-DM1) and Total Trastuzumab - Stage 1
Description: Maximum observed plasma concentration of Trastuzumab Emtansine (T-DM1) and total trastuzumab were reported. Stage 1 consists of all participants recruited before the regimen selection, which was carried out after 12 weeks of randomization.
Time Frame: Day 1 (D1) of Cycle 1 (C1) and C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: Participants who had at least one PK parameter estimated were included for analysis. Here, n=number of participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 41 | 37
microgram per milliliter (mcg/mL)
  T-DM1 Cycle 1 First Dose (n=41, 37) | 43.0 (11.8) | 58.6 (12.9)
  T-DM1 Cycle 4 First Dose (n=25, 10) | 52.6 (19.4) | 61.6 (14.5)
  Total trastuzumab Cycle 1 First Dose (n=41, 37) | 46.8 (12.3) | 61.2 (14.6)
  Total trastuzumab Cycle 4 First Dose (n=25, 10) | 71.2 (23.2) | 66.3 (14.7)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of N2'-Deacetyl-N2'-(3-mercapto-1-oxopropyl)-Maytansine (DM1) - Stage 1
Description: Maximum observed plasma concentration of DM1 were reported. Stage 1 consists of all participants recruited before the regimen selection decision. Regimen selection analysis was carried out after 12 weeks of randomization.
Time Frame: C1D1 and C1C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (mcg/mL)
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 40 | 35
nanogram per milliliter (mcg/mL)
  DM1 Cycle 1 First Dose (n=40, 35) | 2.47 (1.05) | 4.61 (6.26)
  DM1 Cycle 4 First Dose (n=22, 9) | 3.41 (1.61) | 3.86 (0.83)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Trastuzumab Emtansine (T-DM1) and Total Trastuzumab - Stage 2
Description: Stage 2 consists of all participants recruited after the regimen selection decision up to primary data cut-off date 30-June-2015.
Time Frame: C1D1; C4D1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Trastuzumab Emtansine 2.4 mg
Number analyzed (Participants) | 57
mcg/mL
  T-DM1 Cycle 1 First Dose (n=56) | 34.1 (15.2)
  T-DM1 Cycle 4 First Dose (n=26) | 38.0 (13.4)
  Total trastuzumab Cycle 1 First Dose (n=57) | 44.5 (15.4)
  Total trastuzumab Cycle 4 First Dose (n=26) | 69.7 (21.3)

14. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf] - Stage 1
Description: AUCinf= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf). Stage 1 consists of all participants recruited before the regimen selection decision. Regimen selection analysis was carried out after 12 weeks of randomization.
Time Frame: D1C1 and D1C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: Participants who had at least one PK parameter estimated were included for analysis.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 41 | 37
day*mcg/mL
  T-DM1 | 179 (51.0) | 262 (90.3)
  Total trastuzumab | 289 (129) | 403 (237)

15. Secondary Outcome: Plasma Decay Half-Life (t1/2) - Stage 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Stage 1 consists of all participants recruited before the regimen selection decision. Regimen selection analysis was carried out after 12 weeks of randomization.
Time Frame: D1C1 and D1C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: Participants who had at least one PK parameter estimated were included for analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 41 | 37
days
  T-DM1 | 3.48 (0.747) | 3.33 (1.21)
  Total trastuzumab | 5.22 (1.53) | 5.40 (2.15)

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) - Stage 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state. Stage 1 consists of all participants recruited before the regimen selection decision. Regimen selection analysis was carried out after 12 weeks of randomization.
Time Frame: D1C1 and D1C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: Participants who had at least one PK parameter estimated were included for analysis.
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 41 | 37
milliliter per kilogram (mL/kg)
  T-DM1 | 66.2 (19.2) | 67.7 (14.0)
  Total trastuzumab | 65.9 (21.9) | 72.1 (16.1)

17. Secondary Outcome: Systemic Clearance (CL) - Stage 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. Stage 1 consists of all participants recruited before the regimen selection decision. Regimen selection analysis was carried out after 12 weeks of randomization.
Time Frame: D1C1 and D1C4, C1D2, C1D3, C1D4/C1D5, C1D8, C1D15, C2D1 (up to 12 weeks)
Population: Participants who had at least one PK parameter estimated were included for analysis.
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Number analyzed (Participants) | 41 | 37
mL/day/kg
  T-DM1 | 14.6 (4.64) | 15.4 (5.61)
  Total trastuzumab | 10.2 (4.87) | 11.3 (5.46)

ADVERSE EVENTS:
Time Frame: Baseline up to data cut-off date 30-April-2016 (up to 3 years 8 months)
Description: Safety Analysis Population included all participants who received at least one dose of study medication. The safety parameters were analyzed and presented according to the therapy participants received. Cumulative data (up to primary analysis cut-off date of 30-April-2016) are provided for both phase 2 and phase 3.
Arm/Group | Standard Taxane Therapy | Trastuzumab Emtansine 2.4 mg | Trastuzumab Emtansine 3.6 mg
Serious Adverse Events (participants affected / at risk) | 31/111 | 65/224 | 23/69
Other Adverse Events (participants affected / at risk) | 105/111 | 211/224 | 62/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Taxane Therapy (N=111) | Trastuzumab Emtansine 2.4 mg (N=224) | Trastuzumab Emtansine 3.6 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 3 | 8 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 6 | 4
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 5 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 8 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 3
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 7 | 2
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 4 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Taxane Therapy (N=111) | Trastuzumab Emtansine 2.4 mg (N=224) | Trastuzumab Emtansine 3.6 mg (N=69)
Anaemia (Blood and lymphatic system disorders) | 35 | 75 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 10 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 55 | 24 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 60 | 18
Abdominal distension (Gastrointestinal disorders) | 4 | 10 | 6
Abdominal pain (Gastrointestinal disorders) | 12 | 42 | 10
Abdominal pain upper (Gastrointestinal disorders) | 8 | 19 | 6
Constipation (Gastrointestinal disorders) | 22 | 47 | 10
Diarrhoea (Gastrointestinal disorders) | 27 | 33 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 20 | 4
Dyspepsia (Gastrointestinal disorders) | 11 | 17 | 6
Dysphagia (Gastrointestinal disorders) | 4 | 9 | 4
Nausea (Gastrointestinal disorders) | 30 | 57 | 15
Stomatitis (Gastrointestinal disorders) | 21 | 14 | 3
Vomiting (Gastrointestinal disorders) | 15 | 41 | 17
Asthenia (General disorders) | 9 | 39 | 9
Chills (General disorders) | 2 | 12 | 4
Fatigue (General disorders) | 51 | 68 | 24
Malaise (General disorders) | 5 | 12 | 1
Mucosal inflammation (General disorders) | 7 | 8 | 1
Oedema peripheral (General disorders) | 16 | 14 | 5
Pain (General disorders) | 11 | 6 | 3
Pyrexia (General disorders) | 17 | 44 | 11
Alanine aminotransferase increased (Investigations) | 4 | 21 | 5
Aspartate aminotransferase increased (Investigations) | 5 | 36 | 10
Blood alkaline phosphatase increased (Investigations) | 3 | 8 | 5
Blood bilirubin increased (Investigations) | 3 | 13 | 1
Weight decereased (Investigations) | 8 | 13 | 3
Deceased appetite (Metabolism and nutrition disorders) | 32 | 57 | 22
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 13 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 22 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 13 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 13 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 13 | 6
Dizziness (Nervous system disorders) | 5 | 14 | 5
Dysgeusia (Nervous system disorders) | 11 | 18 | 5
Headache (Nervous system disorders) | 6 | 24 | 2
Neuropathy peripheral (Nervous system disorders) | 11 | 22 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 22 | 21 | 4
Depression (Psychiatric disorders) | 0 | 5 | 4
Insominia (Psychiatric disorders) | 10 | 18 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 21 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 57 | 7 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 7 | 4 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 12 | 15 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 26 | 7

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor as the primary analysis results did not meet the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.